CLINICAL TRIAL: NCT01511029
Title: A Single-Center, Randomized, Blinded, Placebo- and Active-Controlled Crossover Study to Evaluate the Effect of Dexpramipexole (BIIB050) on the QTc Interval in Healthy Volunteers
Brief Title: Study to Evaluate the QTC Interval in Healthy Volunteers Dosed With Dexpramipexole (QTC = Electrocardiogram (ECG) Interval Measured From the Onset of the QRS Complex to the End of the T Wave Corrected for Heart Rate)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Knopp Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 223HV102
Record Dates: First submitted 2012-01-09; First posted 2012-01-18 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Dexpramipexole; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dexpramipexole (Experimental)
  Interventions: Drug: Dexpramipexole
- Dexpramipexole (placebo) (Placebo Comparator)
  Interventions: Drug: Dexpramipexole Placebo
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Dexpramipexole — 300 mg - Oral Tablets
  Arms: Dexpramipexole
Drug: Dexpramipexole — 600 mg Oral Tablets
  Arms: Dexpramipexole
Drug: Dexpramipexole Placebo — Placebo - Oral Tablet
  Arms: Dexpramipexole (placebo)
Drug: Moxifloxacin — 400 mg - Oral Tablet
  Arms: Moxifloxacin

SUMMARY:
To evaluate whether dexpramipexole prolongs the QTc interval when orally administered to healthy volunteers.

DETAILED DESCRIPTION:
This is a Phase I, single-center, blinded (with respect to dexpramipexole administration), randomized, placebo- and active-controlled, 4-period crossover study in approximately 68 healthy volunteers. This thorough QT/QTc study will be conducted to formally evaluate the effect of dexpramipexole on QT prolongation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 60 years old inclusive on Day 1.
* Subjects who, in the opinion of the Investigator, are healthy as determined by pre study medical history, physical examination, and 12 lead ECG.
* Male subjects and female subjects of childbearing potential must practice effective contraception (per protocol specifications).
* Normal systemic blood pressure defined as a systolic blood pressure of 90 to 140 mmHg and a diastolic blood pressure of 50 to 90 mmHg.

Exclusion Criteria:

* History of cardiovascular disease (e.g., hypertension, arrhythmia, heart failure, Long QT Syndrome, or other conditions/diseases causing prolongation of the QT/QTc interval), in the opinion of the Investigator.
* A prolongation of QT/QTc interval (e.g., repeated demonstration of a QT/QTc interval >450 ms before study treatment administration.
* Clinically important abnormalities in resting ECG that may interfere with the interpretation of QTc interval changes at screening, check-in, or pre-dose on Day -1 of the first treatment period.
* Other medically significant illness.
* Clinically significant abnormal laboratory values.
* Pregnant women or women breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To evaluate whether a single dose of dexpramipexole prolongs the QTC interval as measured by frequent ECG measurements (using Holter monitoring) of individually corrected QT intervals (QTcI) | change from baseline

SECONDARY OUTCOMES:
Area Under Curve (AUC) of dexpramipexole | pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 23 hours after dosing on Day 1 of each treatment period
Change in ECG measurements | baseline and Day 7
Cmax of dexpramipexole | pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 23 hours after dosing on Day 1 of each treatment period
Tmax of dexpramipexole | pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 23 hours after dosing on Day 1 of each treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Overland Park, Kansas, United States